CLINICAL TRIAL: NCT03063528
Title: Healthy Motivations for Moms-to-be Study
Acronym: HM2B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00061320
Record Dates: First submitted 2017-01-17; First posted 2017-02-24 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Weight Gain; Pregnancy; Stress, Emotional; Exercise; Nutrition
Keywords: Pregnancy; Weight; Gestational weight gain; Stress reduction; Exercise
MeSH Terms: conditions — Weight Gain; Stress, Psychological; Motor Activity; Body Weight; Gestational Weight Gain | interventions — Diet, Healthy; Exercise; Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Healthy Eating/Physical Activity (HEPA) (Experimental): The goals of the HEPA condition are to encourage healthy eating and physical activity behaviors for gaining a healthy amount of weight during pregnancy and to provide motivation and social support to help overcome challenges to eating healthier and becoming more physically active while pregnant.
  * 12 weeks of group-based health behavior (nutrition/PA focused) challenges and weight tracking; podcasts (10); weekly pregnancy tips
  * website and mobile app
  Interventions: Behavioral: Healthy Eating and Physical Activity
- Stress Reduction/Management (SRAM) (Experimental): The goals of the SRAM condition are to encourage stress reduction and management techniques as well as to provide motivation and social support to reduce stress levels during pregnancy.
  * 12 weeks of group-based health behavior (stress reduction/management) challenges and weight tracking; podcasts (10); weekly pregnancy tips
  * website and mobile app
  Interventions: Behavioral: Stress Reduction and Management

INTERVENTIONS:
Behavioral: Healthy Eating and Physical Activity — Participants will be assigned to a group of 8-10 other pregnant women to work towards the same healthy eating or physical activity behavior challenge each week for a total of 12 weeks. The challenges will not require travel or financial support, but will focus on modifying or encouraging daily lifestyle activities, such as "drink 8 full glasses of water 3 times this week." Participants will track their healthy eating and physical activity behaviors in a mobile app. The HEPA condition will have access to podcasts and informational tips for having a healthy pregnancy through the study website. The HEPA condition will be able to log their weight on a daily basis and track their overall weight gain on a chart through the study website.
  Other Names: HEPA
  Arms: Healthy Eating/Physical Activity (HEPA)
Behavioral: Stress Reduction and Management — Participants will be put into a group of 8-10 other pregnant women to work towards the same stress reduction and management goal each week for a total of 12 weeks. The challenges will not require travel or financial support, but will focus on modifying or encouraging daily lifestyle activities, such as "take a 15 minute technology break each day this week." Participants will track their stress reduction and management behaviors in a mobile app. In addition, the SRAM condition will have access to meditation podcasts and informational tips for having a healthy pregnancy through the study website. Lastly, the SRAM condition will be able to rate their stress level on a daily basis and track their stress on a graph.
  Other Names: SRAM
  Arms: Stress Reduction/Management (SRAM)

SUMMARY:
This proposal is part of a broader research agenda that posits healthy gestational weight gain (GWG) may be achieved through behavioral intervention and may potentially reduce adverse maternal and infant health outcomes associated with excessive weight gain during pregnancy. The purpose of this study is to examine the use of a mobile application (mobile app) and mobile website for encouraging and maintaining healthy behaviors such as healthy eating, regular exercise, and stress management and reduction during pregnancy. The study will include collaborative group-based health behavior challenges for pregnant women living in the United States. The study will test the effectiveness of the intervention on improving maternal health behaviors. The proposed research project will examine if an intervention targeting healthy eating and exercise leads to significantly less weight gained during pregnancy versus a comparison group that receives stress reduction and management content.

DETAILED DESCRIPTION:
The purpose of this study is to test the effects of a mobile app and study website for a gestational weight gain intervention targeted to pregnant women living anywhere in the United States (n=130). Participants will be assigned to groups of 8-12 and assigned to two conditions: intervention or comparison. The intervention groups will receive a weight-related intervention (focused on fruit and vegetable intake, self-regulation of foods, and physical activity (PA)), while the comparison groups will receive a non-diet/PA health behavior program (focused on sleep, stress reduction, mental health, and stress management). Participants will be instructed on how to use the a commercially available free mobile app and study website. Each week for 12 consecutive weeks, participants will receive a health related behavioral goal through the mobile app. Participants can track their goal achievements through the app and connect with other pregnant women in the study. The study website will have participants log daily body weight or stress level, based on their respective group assignments. The study website will also offer 10 podcasts and weekly pregnancy tips related to the study content of both groups. Participants will also be asked to complete three online surveys and provide a report of body weight at three time points throughout pregnancy. Participants will receive an incentive gift for their participation.

The proposed research project is significant for several reasons: (1) rates of overweight and obesity among pregnant and postpartum women are increasing, (2) overweight and obesity is associated with unfavorable maternal and child health outcomes and (3) past research has demonstrated the importance of providing social support during pregnancy to reduce antenatal and postpartum depression.

The proposed research project is innovative for several reasons: (1) current modes of delivering interventions are costly and may be limited in reach and scope while mobile technology provides a solution to these burdens, (2) this intervention is the first of its kind to utilize a commercially-available mobile app to address GWG among pregnant women living in the US, (3) using mobile technology for all aspects of the study will allow greater reach to rural populations who have limited ability to regularly receive health information, and (4) this intervention will employ social support strategies by grouping pregnant women into small groups assigned with a weekly weight-related health goal.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant upon enrollment
* Singleton pregnancy
* 20-35 years old
* Current resident of the United States
* Valid email address to receive study updates
* Owner of an Android or iPhone and willing to download a commercially-available, free mobile app

Exclusion Criteria:

* Does not own or cannot access a scale to weigh themselves regularly
* Has uncontrolled/untreated thyroid disease
* Currently takes insulin for diabetes
* Has high blood pressure that is not controlled
* Has had persistent bleeding in the first trimester
* Has a history of 3 or more miscarriages
* Has a history of incompetent (weakened) cervix
* Currently has or has ever had an eating disorder or malnutrition
* Has physical disabilities that prevent her from exercising
* Was told by her doctor that she should NOT exercise during pregnancy

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Total gestational weight gain (kg) | baseline (<20 weeks), 32 weeks, and delivery (40 weeks)
  Photo-verified scale displays at baseline (<20 weeks), 32 weeks, and delivery (40 weeks)

SECONDARY OUTCOMES:
Social engagement within group-based challenges | 12 weeks
  Total engagement score will be computed for app and website usage
Podcast listenership | 20-36 weeks
  Number of podcasts downloaded by individual participant
Motivation to change behavior | baseline (<20 weeks) and 32 weeks
  Surveys administered at baseline (<20 weeks) and 32 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alicia A Dahl, MS, Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://brie.net